CLINICAL TRIAL: NCT05898464
Title: Immunogenicity and Safety of Recombinant Zoster Vaccine in People Living With HIV
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Medical Center, Seoul (Other); SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Wan Beom Park, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2304-110-1426
Record Dates: First submitted 2023-05-30; First posted 2023-06-12 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-03

CONDITIONS: Vaccination; Infection; Vaccine Adverse Reaction
Keywords: Recombinant zoster vaccine; Vaccination of people living with HIV
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HIV #1 (Experimental): CD4+ T cell count <300 cells/µL
  Interventions: Biological: Recombinant zoster vaccination
- HIV #2 (Active Comparator): CD4+ T cell count≥300 cells/µL
  Interventions: Biological: Recombinant zoster vaccination
- non-HIV (Active Comparator): Healthy adult
  Interventions: Biological: Recombinant zoster vaccination

INTERVENTIONS:
Biological: Recombinant zoster vaccination — Two doses of recombinant zoster vaccine(Shingrix®), 2 months apart

SUMMARY:
The purpose of this study is to compare the immunogenicity and safety of recombinant zoster vaccine according to CD4+ T-cell count and age in people living with HIV, and to provide evidence to guide immunization of people living with HIV.

DETAILED DESCRIPTION:
* HIV-infected individuals willing to receive recombinant zoster vaccine will be recruited at three study hospitals.
* Participants are divided into two groups based on HIV status and CD4+ T cell count (HIV #1: CD4+ T cell count <300 cells/µL, HIV #2: CD4+ T cell count≥300 cells/µL, non-HIV).
* Target numbers are 50 for each group.
* Give 2 intramuscular doses of recombinant zoster vaccine 2 months apart.
* Contact by phone on days 3 and 7 after each dose to assess for adverse events.
* Evaluate immunogenicity at 1 month and 13 months after the second dose and safety.
* An interim analysis is planned after the first approximately 30 participants of HIV group and 10 participants of non-HIV group complete a visit 13 months after 2nd dose.
* Evaluation for the safety is planned after the first approximately 10 participants of the HIV #2 arm complete a visit 13 months after 2nd dose.

ELIGIBILITY:
Inclusion Criteria (for HIV #1, HIV #2) :

* 19 years old or older, HIV-1 infected person who have voluntarily agreed to participate in the study.
* Have been taking antiviral medications stably for at least one month at the time of screening.
* Have a CD4+ T-cell count measured before enrollment.
* Do not have AIDS-defining diseases (excluding oral thrush) or acute/uncontrolled opportunistic infection at the time of enrollment.
* Do not have uncontrolled chronic medical conditions other than HIV infection.

Inclusion Criteria (for non-HIV) :

* 50 years old or older who have voluntarily agreed to participate in the study.
* Do not have uncontrolled chronic medical conditions

Exclusion Criteria:

* Have received any type of zoster vaccine within 1 year.
* Have been diagnosed with chickenpox or shingles within 12 months.
* Have a history of severe allergy to any of the components of Shingrix vaccine.
* Have a acute medical condition at the time of screening.
* Unable to be evaluated for adverse events via telephone contact after vaccination.
* Pregnant (including those planning to become pregnant) or lactating women.
* Those who have received chemotherapy or radiotherapy within 6 months prior to the first vaccine dose.
* Chronic administration of immunosuppressive or other immune-modifying drugs within 6 months prior to ther first vaccine dose.
* Administration of immunoglobulins, and/or any blood products within 3 months preceding the first dose of study vaccine
* Have a medical condition that makes receiving an intramuscular injection medically contraindicated.
* Have a disease or condition that may affect the immunogenicity or safety of the vaccine.
* Receiving any other vaccine within 14 days prior to and 14 days after receiving the study vaccine.
* Participate in a clinical trial that involves other investigational product or device during the course of the study.
* Any other person who, in the opinion of the investigator, is unsuitable for immune response assessment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Humoral immune response | 1 month, 13 months after 2nd dose
  Defined as a 4-fold or greater increase in anti-VZV antibody concentration from pre-vaccination testing in seropositive subjects and a 4-fold or greater increase in anti-gE antibody concentration from the cutoff in seronegative subjects prior to vaccination.

SECONDARY OUTCOMES:
Cell-mediated immunogenicity | 1 month, 13 months after 2nd dose
  Defined as a 2-fold or greater increase in CD4+ T cells expressing at least two activation markers (i.e. CD40L, IFN-gamma, IL-2 or TNF-alpha) post-vaccination compared to pre-vaccination baseline.
Differences in humoral immune response and cell mediated immunogenecity | 1 month, 13 months after 2nd dose
  Comparison of geometric mean of anti VZV IgG titer and proportions of VZV-specific CD4+ and CD8+ T-cells between HIV#1 and HIV#2
Grade 3/4 adverse events (AE) | Within 7 days (Day 0-6) after the first and second dose.
  Solicited and unsolicited local and systemic adverse events occurring within 7 days after the first and second dose
Any serious adverse events (SAEs) | Throughout the study period: Day 0~450 or termination, whichever came first
  Any serious adverse events occurring throughout the study period
Increase in HIV Viral Load or decrease in CD4+ T-cell Count | 1 month after 2nd dose
  Increase in HIV Viral Load by 0.5 log or more or decrease in CD4+ T-cell Count by 30% or more
Any AIDS-defining disease | Within 3 months after 2nd dose
  Occurrence of any AIDS defining condition according to the appendix of the "Revised surveillance case definition for HIV infection--United States, 2014" (Centers for Disease Controls and Prevention);

CONTACTS AND LOCATIONS:
Overall Officials: Wan Beom Park, M.D., PhD., Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - National Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No
We are not planning to share IPDs publically, but de-identified individual participant data for all outcome measures could be shared with other researchers under their request.

REFERENCES:
- [Background] Buchbinder SP, Katz MH, Hessol NA, Liu JY, O'Malley PM, Underwood R, Holmberg SD. Herpes zoster and human immunodeficiency virus infection. J Infect Dis. 1992 Nov;166(5):1153-6. doi: 10.1093/infdis/166.5.1153. PMID 1308664
- [Background] Gebo KA, Kalyani R, Moore RD, Polydefkis MJ. The incidence of, risk factors for, and sequelae of herpes zoster among HIV patients in the highly active antiretroviral therapy era. J Acquir Immune Defic Syndr. 2005 Oct 1;40(2):169-74. doi: 10.1097/01.qai.0000178408.62675.b0. PMID 16186734
- [Background] Erdmann NB, Prentice HA, Bansal A, Wiener HW, Burkholder G, Shrestha S, Tang J. Herpes Zoster in Persons Living with HIV-1 Infection: Viremia and Immunological Defects Are Strong Risk Factors in the Era of Combination Antiretroviral Therapy. Front Public Health. 2018 Mar 12;6:70. doi: 10.3389/fpubh.2018.00070. eCollection 2018. PMID 29594092
- [Background] Grabar S, Tattevin P, Selinger-Leneman H, de La Blanchardiere A, de Truchis P, Rabaud C, Rey D, Daneluzzi V, Ferret S, Lascaux AS, Hanslik T, Costagliola D, Launay O; French Hospital Database on HIV (FHDH-ANRS CO4 Cohort). Incidence of herpes zoster in HIV-infected adults in the combined antiretroviral therapy era: results from the FHDH-ANRS CO4 cohort. Clin Infect Dis. 2015 Apr 15;60(8):1269-77. doi: 10.1093/cid/ciu1161. Epub 2015 Jan 18. PMID 25601456
- [Background] Domingo P, Torres OH, Ris J, Vazquez G. Herpes zoster as an immune reconstitution disease after initiation of combination antiretroviral therapy in patients with human immunodeficiency virus type-1 infection. Am J Med. 2001 Jun 1;110(8):605-9. doi: 10.1016/s0002-9343(01)00703-3. PMID 11382367
- [Background] Song JY, Lee JS, Jung HW, Choi HJ, Lee JS, Eom JS, Cheong HJ, Jung MH, Kim WJ. Herpes zoster among HIV-infected patients in the highly active antiretroviral therapy era: Korean HIV cohort study. J Acquir Immune Defic Syndr. 2010 Mar;53(3):417-8. doi: 10.1097/QAI.0b013e3181b1d6dc. No abstract available. PMID 20190589
- [Background] Kim YJ, Woo JH, Kim MJ, Park DW, Song JY, Kim SW, Choi JY, Kim JM, Han SH, Lee JS, Choi BY, Lee JS, Kim SS, Kee MK, Kang MW, Kim SI. Opportunistic diseases among HIV-infected patients: a multicenter-nationwide Korean HIV/AIDS cohort study, 2006 to 2013. Korean J Intern Med. 2016 Sep;31(5):953-60. doi: 10.3904/kjim.2014.322. Epub 2016 Apr 27. PMID 27117317
- [Background] Harbecke R, Cohen JI, Oxman MN. Herpes Zoster Vaccines. J Infect Dis. 2021 Sep 30;224(12 Suppl 2):S429-S442. doi: 10.1093/infdis/jiab387. PMID 34590136
- [Background] Berkowitz EM, Moyle G, Stellbrink HJ, Schurmann D, Kegg S, Stoll M, El Idrissi M, Oostvogels L, Heineman TC; Zoster-015 HZ/su Study Group. Safety and immunogenicity of an adjuvanted herpes zoster subunit candidate vaccine in HIV-infected adults: a phase 1/2a randomized, placebo-controlled study. J Infect Dis. 2015 Apr 15;211(8):1279-87. doi: 10.1093/infdis/jiu606. Epub 2014 Nov 3. PMID 25371534
- [Background] Thompson MA, Horberg MA, Agwu AL, Colasanti JA, Jain MK, Short WR, Singh T, Aberg JA. Primary Care Guidance for Persons With Human Immunodeficiency Virus: 2020 Update by the HIV Medicine Association of the Infectious Diseases Society of America. Clin Infect Dis. 2021 Dec 6;73(11):e3572-e3605. doi: 10.1093/cid/ciaa1391. PMID 33225349
- [Background] Panel on Guidelines for the Prevention and Treatment of Opportunistic Infections in Adults and Adolescents with HIV. Guidelines for the Prevention and Treatment of Opportunistic Infections in Adults and Adolescents with HIV. National Institutes of Health, Centers for Disease Control and Prevention, HIV Medicine Association, and Infectious Diseases Society of America. Available at https://clinicalinfo.hiv.gov/en/guidelines/adult-andadolescent-opportunistic-infection. Accessed March 31, 2023
- [Background] Centers for Disease Control and Prevention (CDC). Revised surveillance case definition for HIV infection--United States, 2014. MMWR Recomm Rep. 2014 Apr 11;63(RR-03):1-10. PMID 24717910